CLINICAL TRIAL: NCT04685694
Title: Expectant Management Versus Medical Management of Retained Products of Conception After Induced Abortion
Brief Title: Management of RPOC After Induced Abortion
Acronym: RPOC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Eli Sprecher, MD, MD, PhD. Deputy Director Research & Development, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0444-19-TLV
Record Dates: First submitted 2020-10-01; First posted 2020-12-28 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Abortion Induced Complicated
Keywords: RPOC, induced abortion, misoprostol
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Expectant (No Intervention): No medication is assigned.
- Medical (Experimental): SL 800 mcg Misoprostol
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — sl 800 mcg misoprostol
  Other Names: Cytotec
  Arms: Medical

SUMMARY:
Randomized trial comparing expectant management and medical management in women diagnosed with retained products of conception after first trimester induced abortion

DETAILED DESCRIPTION:
An open label randomized controlled trial (RCT) of all women diagnosed with retained product of conception (RPOC) after first trimester medical TOP in a single university affiliated medical center. All consecutive women who underwent medical TOP by mifepristone and misoprostol at gestational age under 63 days from last menstrual period and were diagnosed with RPOC in a routine 3-week ultrasound follow-up are offered to participate. RPOC is defined as thick irregular endometrium (over 12 mm) with positive Doppler flow. Following recruitment, patients are randomized into either expectant arm or medical arm (800 mcg misoprostol). The primary outcome measure is RPOC rate in repeat ultrasound scan performed 5 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

* 18 < age < 45 year old
* Thick irregular endometrium >12 mm on trans-vaginal ultrasound

Exclusion Criteria:

* Endometritis
* Cervical opening > 1 cm
* Uterine abnormalities
* Contraindication to Misoprostol treatment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
RPOC rate | 2 months
  RPOC rate in repeat ultrasound scan performed 5 weeks after randomization

SECONDARY OUTCOMES:
Adhesions | 2 months
  According to our study protocol all women with persistent products of conception diagnosed on repeated ultrasound examination undergo hysteroscopy. During hysteroscopy, assessment of the uterine cavity including intrauterine adhesion formation will be performed. Intrauterine adhesions will be classified according to the American Society for Reproductive Medicine (ASRM), based on the extent of cavity involvement (<1/3; 1/3 to 2/3, >2/3) and the type of adhesion seen (filmy, filmy and dense, dense).
Bleeding | 2 months
  Bleeding pattern will be assessed via questionnaire upon recruitment and follow up visits. Bleeding will be characterized by its pattern (regular, intermenstrual) and quantity (normal, hypomenorrhoea, menorrhagia).

CONTACTS AND LOCATIONS:
Overall Officials: Yossi Tzur, MD, Study Director — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center; ,, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
on line sharing via secured system
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years
Access Criteria: for research purposes only

REFERENCES:
- [Background] Trinder J, Brocklehurst P, Porter R, Read M, Vyas S, Smith L. Management of miscarriage: expectant, medical, or surgical? Results of randomised controlled trial (miscarriage treatment (MIST) trial). BMJ. 2006 May 27;332(7552):1235-40. doi: 10.1136/bmj.38828.593125.55. Epub 2006 May 17. PMID 16707509
- [Background] Bagratee JS, Khullar V, Regan L, Moodley J, Kagoro H. A randomized controlled trial comparing medical and expectant management of first trimester miscarriage. Hum Reprod. 2004 Feb;19(2):266-71. doi: 10.1093/humrep/deh049. PMID 14747165
- [Background] Ashwal E, Melamed N, Hiersch L, Wiznitzer A, Yogev Y, Peled Y. The incidence and risk factors for retained placenta after vaginal delivery - a single center experience. J Matern Fetal Neonatal Med. 2014 Dec;27(18):1897-900. doi: 10.3109/14767058.2014.883374. Epub 2014 Feb 4. PMID 24417417
- [Background] Anteby M, Many A, Ashwal E, Yogev Y, Shinar S. Risk factors and complications of manual placental removal after vaginal delivery - how common are additional invasive procedures? J Matern Fetal Neonatal Med. 2019 Feb;32(3):384-388. doi: 10.1080/14767058.2017.1379071. Epub 2017 Sep 19. PMID 28891361
- [Derived] Tzur Y, Berkovitz-Shperling R, Goitein Inbar T, Bar-On S, Gil Y, Levin I, Cohen A. Expectant vs medical management for retained products of conception after medical termination of pregnancy: a randomized controlled study. Am J Obstet Gynecol. 2022 Oct;227(4):599.e1-599.e9. doi: 10.1016/j.ajog.2022.06.025. Epub 2022 Jun 23. PMID 35752301